CLINICAL TRIAL: NCT00523458
Title: A Study to Determine the Best Dose of Antivirals in Patients With Both TB and HIV
Acronym: OPTI-NNRTI
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: A delay in protocol approval and approval of laboratory sites in Salvador, Brazil left too little time for completion of enrollment into the study.
Sponsor: Stanford University (Other)
Responsible Party: Terrence F Blaschke, Principle Investigator, Stanford University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Stanford Protocol ID: 95564
Record Dates: First submitted 2007-08-29; First posted 2007-08-31 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: HIV Infections; Tuberculosis
Keywords: Co-infection; Tuberculosis; HIV; Drug interactions; Non nucleoside reverse transcriptase inhibitors; Therapy; Treatment Naive
MeSH Terms: conditions — HIV Infections; Tuberculosis; Coinfection | interventions — efavirenz; Nevirapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): Standard dose nevirapine (200 mg 2x daily) in combination with 2 nucleoside analogs
  Interventions: Drug: efavirenz or nevirapine
- 2 (Experimental): High dose nevirapine (400 mg in the morning, 200 mg in the evening) in combination with 2 nucleoside analogs
  Interventions: Drug: efavirenz or nevirapine
- 3 (Active Comparator): Standard dose efavirenz (600 mg at bedtime) in combination with 2 nucleoside analogs
  Interventions: Drug: efavirenz or nevirapine
- 4 (Experimental): High dose efavirenz (800 mg at bedtime) in combination with 2 nucleoside analogs
  Interventions: Drug: efavirenz or nevirapine

INTERVENTIONS:
Drug: efavirenz or nevirapine — Patients co-infected with HIV and TB will receive either "standard" doses of nevirapine (200 mg 2x daily) or efavirenz (600 mg daily) or "high" doses of nevirapine (400 mg and 200 mg daily) or efavirenz (800 mg daily) that are chosen to compensate for the change in pharmacokinetics shown to occur when co-infected patients are treated with the antituberculous drug, rifampin.
  Other Names: Sustiva (efavirenz); Viramune (nevirapine)

SUMMARY:
Because drugs used to treat TB can reduce the amount of the anti-HIV drugs that reach the sites where the virus is located, this study is designed to see whether it is necessary to use higher doses of antiviral (anti-HIV) drugs while patients are receiving therapy with rifampin, one of the drugs commonly used to treat TB. Participants will be assigned to one of 4 arms (see below) and will be followed during the time when they are receiving both treatments.

DETAILED DESCRIPTION:
This is an open label, randomized study with 4 arms: 1.) Standard dose and 2.) high dose nevirapine; and 3.) standard dose and 4.) high dose efavirenz. Subjects in all 4 arms will also receive 2 nucleoside analog drugs. Patients will have routine monitoring for the treatment of TB and HIV, as well as some additional blood samples to follow the virus in the blood and to determine the effect of the TB therapy on the amounts of anti-HIV drugs that are in the body.

ELIGIBILITY:
Inclusion Criteria:

* ARV naïve subjects
* Documented HIV infection
* Documented TB infection
* Platelet count 40,000/mm3
* Hemoglobin ≥8.0 g/dL
* Absolute neutrophil count (ANC) >500/mm3
* AST (SGOT), ALT (SGPT), and alkaline phosphatase <3 X ULN
* Total bilirubin <2.5 x ULN
* Calculated creatinine clearance ≥60 mL/min
* For women of reproductive potential, negative urine pregnancy test

Exclusion Criteria:

* Unable to provide informed consent.
* History drug abuse that the investigators suspect will interfere with compliance to study medications and visits.
* Patients on hemodialysis.
* Tuberculosis meningitis.
* Women with CD4 > 250 and men with CD4 > 400 due to higher risk of hepatotoxicity related to use of NVP.
* Positive serology for hepatitis C.
* Evidence for active hepatitis B including positive serologies for HBsAg, HBeAg, or HBV-DNA. Note: If anti-HBs is positive, patient is eligible for study if liver enzymes are within the parameters indicated in the inclusion criteria
* Women who are breast-feeding
* Known allergy/sensitivity to study drug(s) or their formulations
* Patients with other OIs or intercurrent illness that could affect their ability to take study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-07; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Decline in HIV RNA in plasma Rise in CD4 cell count | Baseline, and Weeks 8, 20 and 32
  These laboratory measures would be used to determine if there was a difference in the ARV failure rate between patients receiving standard dose vs high dose treatment with NNRTIs

CONTACTS AND LOCATIONS:
Overall Officials: Terrence F Blaschke, M.D., Principal Investigator — Stanford University
Locations (1):
- Hospital Universitario Prof. Edgard Santos/Universidade Federal da Bahia, Salvador, Estado de Bahia, Brazil